CLINICAL TRIAL: NCT06262308
Title: Emotional Support for Women Experiencing Preterm Prelabour Rupture of the Membranes (PPROM) - a Research Study
Brief Title: Emotional Support for Women Experiencing PPROM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 334235
Record Dates: First submitted 2024-02-01; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Fetal Membranes, Premature Rupture; Preterm Birth Complication
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Intervention Model Description: This is a pilot study where a small cohort of women will give given personalised psychological intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychological intervention (Experimental): Women will be given psychological intervention
  Interventions: Behavioral: Psychological intervention along Cognitive Behavioural Therapy principles

INTERVENTIONS:
Behavioral: Psychological intervention along Cognitive Behavioural Therapy principles — Women who have PPROM will be offered a series of 6 sessions with a Clinical Psychologist

SUMMARY:
Preterm Prelabour Rupture of the Membranes is a pregnancy complication affecting 3% of all pregnancies. Outcomes for both the mother and baby are variable including: preterm delivery, fetal infection, cord prolapse, abruption as well as maternal sepsis and even maternal death. The outcomes are not only variable but the stress and uncertainty can be over a protracted period of time. This is a pilot study that aims to provide personalised psychological intervention at the time of PPROM based on Cognitive Behavioural Principles to see whether this improves psychological outcomes for women.

DETAILED DESCRIPTION:
Preterm Prelabour Rupture of Membranes PPROM affects 3% of all pregnancies. Outcome is variable depending on the time the waters break. Complications include preterm delivery, infection for both mother and baby, umbilical cord prolapse and abruption. In addition if the membranes rupture before 24 weeks women are offered termination of pregnancy due to the risk of pulmonary hypoplasia (underdeveloped lungs). If infection is not present and labour does not occur delivery may be deferred until 37 weeks. Consequently the condition can be associated with prolonged periods of psychological uncertainty.

There is good evidence to suggest that psychological support at the time of traumatic events reduces the long term psychological consequences ie post traumatic stress disorder. Although national guidelines on PPROM suggest psychological support should be available this is not routine clinical practice and no guidance is given on what form of support this should be.

This pilot study aims to develop a talking therapy based on Cognitive Behavioural Therapy principles to support women and garner their feedback.

A series of 5-8 women who are hospitalised in St Thomas' hospital where their waters have broken before 37 weeks into their pregnancy will be approached by a member of the team of doctors/midwives who are looking after them.

Women will be offered an initial session of assessment by a psychologist to gain an individualised understanding of their current anxiety and mood levels and to assess what is causing stress. This may be thoughts, feelings and behaviours relative to their current mood and aspects of the current situation. A set of strategies will be developed such as education about anxiety and responses to traumatic and upsetting situations, modification of negative thoughts, support with excessive reassurance seeking, self-compassionate exercises to help with self-criticism and self-blame, support with decision-making and strategies to manage uncertainty.

Up to 5 further hour long follow up sessions will occur with the time between sessions and number determined by the woman and her circumstances. Due to the levels of uncertainty associated with the situation, each session will be considered as a stand-alone.

Information about their details (such as age, ethnicity, whether they currently have a partner, details of medical conditions, current and previous pregnancies) will be obtained from participants. A brief measure of mood will be collected at each contact and at 4-6 weeks after the final session. The Hospital Anxiety and Depression scale a validated tool will be used to assess mood.

Given that women will be in the midst of a potentially fast-moving medical context may affect scores to some extent, further feedback will be sought from women at the end of each therapy session and beginning of each subsequent session on how useful they have found the session and interventions suggested.

Detailed notes will be kept on the specific techniques employed in each session and suggested as between session practice.

ELIGIBILITY:
Inclusion Criteria:

* Woman (or birthing person) aged 16 years or over;
* Is experiencing PPROM
* Has been admitted to the ward
* Has capacity to give informed consent to take part in the research
* Speaks and writes English

Exclusion Criteria:

• Unable or unwilling to give informed consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women or individuals who are pregnant
Enrollment: 8 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Mood Score 1 | Through study on average 3 months
  The Depression Anxiety Stress Scale 21 (a set of three self reported scales measuring depression anxiety and stress the higher the score the worse the symptoms. For depression 28+ is extremely severe, for anxiety 20+ is extremely severe and 34+ is extremely severe stress).
Mood Score 2 | Through study on average 3 months
  Based on the Hospital Anxiety and Depression Scale (this encompasses seven questions scored separately for anxiety and depression, 8-10 is mild, 11-14 is moderate and 15-21 is severe for anxiety/depression)
Participant Feedback | Through study and on completion of the study: on average eight months
  Feedback will be sought from participants. This will encompass free text on how useful they felt the sessions had been. A Likert scale will also be incorporated into this questionnaire: score 0-10 (0 not useful, 10 extremely useful).

CONTACTS AND LOCATIONS:
Locations (1):
- St Thomas' Hospital, King's College London, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is a pilot study only but data will be shared with academic institutions on request